CLINICAL TRIAL: NCT05881681
Title: A Mindfulness Approach to Unwinding Anxiety for Afro-descendants
Brief Title: A Mindfulness Approach to UA for Afro-descendants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Richard King Mellon Foundation (Unknown); University of Pittsburgh Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2112003165
Record Dates: First submitted 2022-11-04; First posted 2023-05-31 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Anxiety; Stress
Keywords: Worry
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App-Delivered Mindfulness Training (MT) (Experimental): The Unwinding Anxiety program is delivered via a smartphone-based platform, which includes a progression through 30+ daily modules of brief didactic and experience-based mindfulness training (videos and animations), app-triggered check-ins to encourage engagement, and user-initiated guided mindfulness exercises to help disrupt worry cycles in the moment.
  Interventions: Behavioral: App-Delivered Mindfulness Training (MT)

INTERVENTIONS:
Behavioral: App-Delivered Mindfulness Training (MT) — Unwinding Anxiety is an app-delivered mindfulness training program which includes a progression through 30+ daily modules. Each module's training is delivered via short video tutorials and animations (~10 min/day). Each training builds on the previous one; modules are 'locked' so that they can only be viewed at a pace of 1/day (previous modules can be reviewed at any time). A built-in self-assessment is taken after every seven modules to ensure key concepts are learned before moving on with automated suggestions on which modules to repeat based on the self-assessment results. User-initiated guided practices range from short exercises (30 seconds) to manage anxiety the moment it arises to formal guided meditations (up to 15 minutes), and can be accessed at any time

SUMMARY:
The goal of this clinical trial is to test an app-based mindfulness training program in an Afro-descendant population. The main question[s] it aims to answer are:

* What changes, if any, does the app need?
* Is it effective in reducing anxiety among this population?

Participants will be asked to:

* Use an app-based mindfulness training program daily
* Complete online surveys at baseline and 2 months post-treatment initiation
* Complete focused interviews via Zoom at baseline and 2 months post-treatment initiation
* Complete daily voice diaries via Zoom

ELIGIBILITY:
Inclusion Criteria:

* GAD-7 ≥ 10
* Self-identify as Black American and/or Afro-descendant
* Located in United States or Canada
* Able to speak English
* Owns a smartphone

Exclusion Criteria:

* Any usage of psychotropic medication: not on a stable dosage 6+ weeks
* As needed (i.e., prn) benzodiazepine use
* Psychotic disorder (e.g., bipolar disorder, schizophrenia, schizoaffective disorder, psychosis)
* Cohabiting with a study participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Focused interviews | Baseline
  In-depth interviews will be conducted to collect participant feedback.
Focused interviews | 2 months
  In-depth interviews will be conducted to collect participant feedback.

SECONDARY OUTCOMES:
Change in anxiety | Baseline, 2 months
  Generalized Anxiety Disorder 7-item will be used to assess anxiety. The GAD-7 is a 7-item questionnaire that uses a 4-point Likert scale where 0 is "Not at all" and 3 is "Nearly every day". Scores can range from 0 to 21 and higher scores indicated a worse outcome.
Change in worry | Baseline, 2 months
  Penn State Worry Questionnaire (PSWQ) will be used to assess worry. The PSWQ is a 16-item questionnaire that uses a 5-point Likert scale where 1 is "Not at all typical of me" and 5 is "Very typical of me". Scores can range from 16 to 80 and higher scores indicate a worse outcome
Change in non-reactivity | Baseline, 2 months
  Non-reactivity subscale from the 15-item Five Facet Mindfulness Questionnaire (FFMQ) will be used to measure changes in emotional reactivity. This subscale is based on responses to 3 questions measured on a 5-point Likert scale where 1 is "Never or rarely" and 5 is "Very often or always true". Scores can range from 3 to 15 and higher scores indicate a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Judson A Brewer, Principal Investigator — Brown University
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No